CLINICAL TRIAL: NCT00873340
Title: Physical Disability Observational Study in Patients Treated With Betaferon in Daily Practice
Brief Title: Physical Disability in Patients Treated With Betaferon
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 14173; BF0712CO (Other: company internal); 2007- 001 Col (Other: company internal)
Record Dates: First submitted 2009-03-31; First posted 2009-04-01 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Multiple Sclerosis
Keywords: MS; Multiple Sclerosis; Betaferon; Colombia
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1b

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Interferon-1beta (Betaseron, BAY86-5046)

INTERVENTIONS:
Drug: Interferon-1beta (Betaseron, BAY86-5046) — Patients with a first demyelinating event suggestive of MS, as well as patients with remittent recurrent MS (RRMS), secondary progressive MS (SPMS) and primary progressive MS (PPMS) will be observed.

SUMMARY:
To gather Observation data about physical disability progression, safety and adherence during the use of Betaferon in daily practice. Patients with any type of Multiple Sclerosis (MS) (MRRS) (PSMS), under treatment with Betaferon.Open Multicentric Observational study.24 months.Evaluation of physical disability in patients treated with Betaferon, using Kurtzke's expanded disability scale (EDSS) in biannual periods

ELIGIBILITY:
Inclusion Criteria:

* Patients with a first demyelinating event suggestive of MS, as well as patients with remittent recurrent MS (RRMS), secondary progressive MS (SPMS) and primary progressive MS (PPMS) will be able to join the study.

Exclusion Criteria:

* Pregnancy
* Patients with a history of hypersensitivity to natural or recombinant interferon-beta, human albumin or to any of the excipients
* Patients with a history of severe depressive disorders and/or suicidal ideation
* Patient with decompensated liver disease
* Patient with epilepsy not adequately controlled by treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MS community sample
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2007-10; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
To collect observational local data about effectivity related to physical disability progression on the daily routine basis in patients treated with Betaferon | Every 6 months for 2 years

SECONDARY OUTCOMES:
To evaluate Betaferon safety on the daily routine basis | Every 6 months
To evaluate patient adherence to Betaferon treatment | Every 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Colombia